CLINICAL TRIAL: NCT04085406
Title: Deep Brain Stimulation of the Subgenual Cingulate Cortex for the Treatment of Medically Refractory Chronic Low Back Pain
Brief Title: DBS of the SCC for the Treatment of Medically Refractory CLBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Ausaf A. Bari, MD, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UH3NS113661 (NIH); UH3NS113661 (NIH)
Record Dates: First submitted 2019-08-30; First posted 2019-09-11 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Stimulation (Experimental): Patients will be randomized in a 1:1 ratio to one of two groups: Active Treatment (active stimulation programmed to the settings found to be optimal during the initial open-label period) and a Control Group (sham stimulation - IPG is set to ON but the voltage is set to 0V).
  Interventions: Device: Deep Brain Stimulation of the Subgenus Cingulate Cortex
- Sham Stimulation (Sham Comparator): Patients will be randomized in a 1:1 ratio to one of two groups: Active Treatment (active stimulation programmed to the settings found to be optimal during the initial open-label phase) and a Control Group (sham stimulation - IPG is set to ON but the voltage is set to 0V).
  Interventions: Device: Deep Brain Stimulation of the Subgenus Cingulate Cortex

INTERVENTIONS:
Device: Deep Brain Stimulation of the Subgenus Cingulate Cortex — The Abbott Infinity DBS device will be surgically implanted in the bilateral subgenual cingulate cortex to provide electrical stimulation to this region.

SUMMARY:
The purpose of this study is to evaluate the feasibility and preliminary efficacy of deep brain stimulation of the subgenual cingulate cortex for the treatment of chronic medically-refractory low back pain using a randomized double-blind crossover design.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is one of the most ubiquitous and intractable problems in medicine and a significant source of patient suffering and disability, leading to opioid misuse and addiction. Previous neuromodulatory therapies for CLBP have focused primarily on spinal etiologies and intra-spinal mechanisms of pain transmission. However, existing pharmacological and neuromodulatory therapies have not been successful in treating CLBP. This project aims to address critical gaps and the unmet therapeutic needs of CLBP patients by using the Abbott Infinity DBS System; a next generation DBS device with directional steering capability implanted bilaterally in the subgenual cingulate cortex (SCC) to engage networks known to mediate the affective component of CLBP. The objective is to (1) Assess the preliminary efficacy of DBS of the SCC in the treatment of medically refractory CLBP; (2) Demonstrate the safety and feasibility of SCC DBS for CLBP; and (3) Develop diffusion tensor imaging (DTI)-based blueprints of response to SCC DBS for CLBP. The overall impact of this proof-of-concept pilot trial includes validation of the concept that suffering from CLBP results from pathological activity in affective brain networks, that these networks can be accurately engaged using a next-generation directional DBS device in a safe and feasible manner, and the discover of neuroimaging biomarkers of response to SCC DBS for CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Pain secondary to failed back surgery syndrome (FBSS) as defined by persistent low back pain despite prior surgical interventions.
* Self-reported average back pain intensity of greater than 8 out of 10 on the Visual Analog Scale (VAS) documented over greater than 2 years.
* Failure to achieve at least 50% pain relief from a trial of spinal cord stimulation (SCS) or less than 50% pain relief after 3 months of SCS therapy or patient refuses/rejects SCS trial
* Failure to achieve at least 50% pain relief in response to at least 4 weeks of physical therapy.
* Failure to achieve at least 50% pain relief in response to at least 2 percutaneous spinal pain procedures.
* Failure to achieve at least 50% pain relief in response to 3 months of opioid therapy (at least 20 MEQ/day) or inability to increase or tolerate opioid therapy due to dose-limiting side effects).
* Failure to achieve at least 50% pain relief in response to a 3-month trial of at least one other class of pain medication in addition to opioid therapy or inability to tolerate increasing doses of non-opioid pain medications due to dose-limiting side effects.
* Lack of a surgically correctible etiology for the pain as determined by 2 independent neurosurgeons
* Age greater than 40 years of age.
* Ability to give informed consent in accordance with institutional policies and participate in the 1.5-year follow-up, involving assessments and stimulator adjustments.
* Willingness to share unexpected neurological or psychiatric symptoms with study clinicians.

Exclusion Criteria:

* Significant neurocognitive impairment (MoCA < 26).
* Age > 75 years.
* History of implant-related infection.
* History of bleeding disorder or immune-compromise.
* Psychiatric comorbidity other than depression or generalized anxiety disorder, as determined by MINI International Neuropsychiatric Interview.
* Patients with neurological diagnoses that may reduce the response to or increase the risk of DBS including neurodegenerative conditions, severe movement disorders, demyelinating disorders, syringomyelia, epilepsy or history of seizures, history of CNS tumors (spinal and/or cranial), history of serious head injury with loss of consciousness, history of stroke, surgically reversible peripheral pain syndromes including surgically correctable radiculopathy, and severe peripheral neuropathy.
* Patients who have undergone spine surgery within the previous 3 months.
* Major medical co-morbidities increasing the risk of surgery including uncontrolled hypertension, severe diabetes, major organ system failure, history of hemorrhagic stroke, need for chronic anticoagulation, active infection, immunocompromised state or malignancy with < 5 years life expectancy.
* Individuals with a currently implanted SCS device.
* Individuals with a life expectancy less than 1 year due to any cause.
* Individuals involved in an injury claim under current litigation.
* Individuals with a pending or approved worker's compensation claim.
* Patient living greater than 100 miles from UCLA.
* Suicide attempt in the last two years and/or presence of a suicide plan (an answer of Yes to Question C4 in Section C- Suicidality of MINI International Neuropsychiatric Interview).
* Alcohol or illicit substance use disorder (other than nicotine) within the last 6 months, unstable remission of substance abuse, or chart evidence that co-morbid substance use disorder could account for lack of treatment response.
* Uncontrolled medical condition including cardiovascular problems and diabetes.
* Pregnant or planning to become pregnant.
* Use of warfarin or other blood thinners.
* Significant structural abnormality on preoperative brain MRI.
* Contraindications to MRIs or the need for recurrent body MRIs.
* Presence of cardiac pacemakers/defibrillators, implanted medication pumps, intra-cardiac lines, any intracranial implants (e.g., aneurysm clip, shunt, cochlear implant, electrodes) or other implanted stimulators.
* History of prior cranial neurosurgery.
* Patients unable to discontinue any existing therapeutic diathermy.
* Individuals who are concomitantly participating in another clinical study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of at least 50% in pain scores on the visual analog scale (VAS) compared to baseline. | 12 months - the end of the crossover period
  The visual analog scale for pain is a continuous horizontal scale of length 100 mm with the extremes of pain expressed on either end (0 = no pain, 10 = worst pain). The change on the VAS from active stimulation compared to baseline and sham stimulation will be calculated.
Change in at least 50% in pain scores on the Pain Anxiety Symptoms Scale -- Short Form 20 (PASS SF-20) compared to baseline. | 12 months - the end of the crossover period
  The PASS SF-20 score is a composite 20 item score which focuses on fear and anxiety of pain. It includes 4 sections on aspects of pain including cognitive, escape/avoidance, fear and physiological anxiety. All items are rated on a scale from 0 (never) to 5 (always), where higher values indicate worse outcome. Summary scores are calculated by summing assigned items and then by summing the subscales to derive an overall score for a possible total of 100. The change on the PASS from active stimulation compared to baseline and sham stimulation will be calculated.
At least 10% of study participants to experience one or more significant adverse events (SAEs) | 18 months - the end of the study
  The percentage of subjects with one or more SAEs during the entire study period will be calculated.

SECONDARY OUTCOMES:
Change in dose and/or frequency of opioid analgesic medication use in oral morphine equivalents. | 12 months - the end of the crossover period
  The effect of therapy on reduction in opioid medication intake will be compared to baseline. Opioid use will be converted into morphine milligram equivalents (MME). The MME taken in the preceding month will be calculated using chart review and expressed in MMEs/ day and total MMEs/month expressed as a percentage of the baseline usage calculated as the average MMEs/day and MMEs/month over the previous six months before the start of enrollment. The change from active stimulation compared to baseline and sham stimulation will be calculated.
50% improvement in McGill Pain Questionnaire (MPQ) | 12 months - the end of the crossover period
  The McGill Pain Questionnaire (MPQ) is a well validated and reliable measure of pain. The MPQ captures pain intensity on a 0 to 10 scale where 0 is no pain and 10 is pain as bad as it can be. It is a well validated measure of sensory, affective, and evaluative pain.
Change in Short-Form 36 (SF-36) quality of life questionnaire score. | 12 months - the end of the crossover period
  Short Form 36. The SF-36 Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used in health economics as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in EuroQol 5-Domain (EQ-5D) Score | 12 months - the end of the crossover period
  The EQ-5D is a 5-item patient self-reported survey of health-related quality of life questions consisting of a descriptive part and an evaluation part. The descriptive part includes 5 categories: mobility, self-care, usual activities, pain/ discomfort, and anxiety/depression. Each category can be rated as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3 - for a total of the 5 categories. In the evaluation part, subjects rate their overall health on a visual analog scale (0 to100, where 100 is most healthy). The change in the EQ-5D score from active stimulation compared to baseline and sham stimulation will be calculated.
Change in Montreal Cognitive Assessment Score (MoCA) | 12 months - the end of the crossover period
  The MoCA is a 30-point cognitive test which measures memory, visuospatial ability, executive function, attention, language and orientation to time and place. The MoCA score will be used to assess potential adverse effects of stimulation on cognition. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal. The change in the MoCA score from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the Hamilton Depression Rating Scale (HAM-D) | 12 months - the end of the crossover period
  The HAM-D is a 17-item rating scale for depression. It is the most frequently used depression rating scale used in controlled clinical trials. It provides ratings on current DSM-IV symptoms of depression, with the exceptions of hypersomnia, increased appetite, and concentration/indecision. The HAMD-17 was designed to be administered by a trained clinician using a semi-structured clinical interview. The 17- items are rated on either a 5-point (0-4) or a 3-point (0-2) scale.The change in the HAM-D score from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the Oswestry Disability Index (ODI) | 12 months - the end of the crossover period
  The ODI is a self-assessment of disability secondary to low back pain. The ODI consists of ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each item is rated from 0 to 5, the item scores summed and then multiplied by 2 to arrive at a combined final index score ranging from 0 (no disability) to 100 (highest disability),. The change in the ODI from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the NIH Toolbox Pain Interference Computer Adaptive Test (CAT) | 12 months - the end of the crossover period
  NIH Toolbox Pain Interference CAT asks participants about how their experience of pain interfered with or affected their enjoyment of various daily activities in the past seven days. The CAT scale is computer-adaptive and has a minimum of four questions and a maximum of 12 questions. The questions ask for a response on a 5-point scale: "Not at all" to "Very much"; or rated: "Never" "Always". The test is self-assessed using the NIH Toolbox app which will be installed on an iPad provided to the subject for the duration of the study. The survey is scored using IRT (item response theory) methods. An IRT theta score is generated for each participant, and while no Toolbox norms are available for this measure, the IRT scores are converted to general T-scores based off PROMIS (pain intensity scale). Higher theta and T-Scores represent greater participant report of pain interference. The change from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the PROMIS Pain Intensity Scale 3a | 12 months - the end of the crossover period
  PROMIS Pain Intensity Scale 3a fixed form test consists 3 questions about the subject's worst pain and average pain over the past 7 days and current pain level. All items are self-reported on a scale of 1 (no pain) -5 (maximal pain). The test is self-assessed using the NIH Toolbox app which will be installed on an iPad provided to the subject for the duration of the study. The change from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the PROMIS Pain Behavior CAT | 12 months - the end of the crossover period
  The PROMIS Pain Behavior CAT measures pain related behavioral changes. All items are self-reported on using the NIH Toolbox app which will be installed on an iPad provided to the subject for the duration of the study. With CAT, participant responses guide the system's choice of subsequent items from the full item bank (20 items in total). The score metric is Item Response Theory (IRT), a family of statistical models that link individual questions to a presumed underlying trait or concept of pain behavior represented by all items in the item bank. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. The change from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the NIH Toolbox Positive Affect CAT | 12 months - the end of the crossover period
  The NIH Toolbox Positive Affect CAT measures positive affect. All items are self-reported on using the NIH Toolbox app which will be installed on an iPad provided to the subject for the duration of the study. The score metric is Item Response Theory (IRT). The change from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the NIH Toolbox Sadness CAT | 12 months - the end of the crossover period
  The NIH Toolbox Sadness CAT measures the subject's level of sadness. All items are self-reported on using the NIH Toolbox app which will be installed on an iPad provided to the subject for the duration of the study. The score metric is Item Response Theory (IRT). The change from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the NIH Toolbox General Life Satisfaction CAT | 12 months - the end of the crossover period
  The NIH Toolbox General Life Satisfaction CAT measures life satisfaction. All items are self-reported on using the NIH Toolbox app which will be installed on an iPad provided to the subject for the duration of the study.The score metric is Item Response Theory (IRT). The change from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the NIH Toolbox Perceived Stress Fixed Form (FF) | 12 months - the end of the crossover period
  The NIH Toolbox Perceived Stress FF is a 10-item measure of perceived stress. All items are selfreported on using the NIH Toolbox app which will be installed on an iPad provided to the subject for the duration of the study. The score metric is Item Response Theory (IRT). The change from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the PROMIS Prescription Pain Medication Misuse CAT | 12 months - the end of the crossover period
  The PROMIS Prescription Pain Medication Misuse CAT is a 17-item measure of misuse and/or abuse of prescription pain medications. All items are self-reported on using the NIH Toolbox app which will be installed on an iPad provided to the subject for the duration of the study. The score metric is Item Response Theory (IRT). The change from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the NIH Toolbox Locomotion | 12 months - the end of the crossover period
  The NIH Toolbox Locomotion measures locomotion. Participants walk a short distance at their usual pace, completing one practice and two-timed trials. Scores are recorded as time in seconds required to walk 4 meters on each of two trials, with the better trial used for scoring. An administrator will use the NIH toolbox app to assist in conducting this assessment. The change from active stimulation compared to baseline and sham stimulation will be calculated.
Change in the NIH Pain Intensity Survey | 12 months - the end of the crossover period
  NIH Toolbox Pain Intensity Survey consists of one self-report item asking about the participant's level of pain in the past seven days. Participants are asked to rate their pain on a scale from 0 (no pain) to 10 (worst imaginable pain). All items are selfreported on using the NIH Toolbox app which will be installed on an iPad provided to the subject for the duration of the study. The change from active stimulation compared to baseline and sham stimulation will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ausaf Bari, MD PhD, Principal Investigator — UCLA Department of Neurosurgery
Locations (2):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No